CLINICAL TRIAL: NCT05263765
Title: Aortic Occlusion for Resuscitation in Trauma and Acute Care Surgery (AORTA)
Brief Title: Aortic Occlusion for Resuscitation in Trauma and Acute Care Surgery
Status: Enrolling by invitation | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 063.TRA.2021.D
Record Dates: First submitted 2022-02-03; First posted 2022-03-03 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Aortic Occlusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: utilization of AO in the acute resuscitation of trauma and acute care surgery patients in shock. — AO to facilitate the acute resuscitation of trauma and acute care surgery patients in shock.

SUMMARY:
Aortic occlusion (AO) for trauma has traditionally been accomplished by supra-diaphragmatic clamping of the descending thoracic aorta via emergent thoracotomy or as an initial step during laparotomy.

DETAILED DESCRIPTION:
An evolution in endovascular technologies, however, has provided additional means by which to achieve AO. Expanding experience with the utilization of balloon occlusion in the setting of abdominal aortic rupture due to chronic vascular disease has demonstrated the potential of these new technologies. Discussion of the employment of endovascular AO in the realm of trauma has led to the description of this approach and the demonstration of its effectiveness in animal models of severe hemorrhage.

The purpose of the present study is to prospectively examine the modern utilization of AO in the acute resuscitation of trauma and acute care surgery patients in shock.

ELIGIBILITY:
Inclusion Criteria:

* All adult (age ≥ 18 years) trauma and acute care surgery patients treated with resuscitative AO (via open or endovascular means) in the acute phases after injury
* Transient or refractory hypotension (systolic blood pressure <90mmHg) with a positive abdominal focused abdominal sonography in trauma (FAST) scan, severe pelvic fracture(s), or neither with persistent hypotension without obvious source
* Chest x-ray without evidence of thoracic aortic injury
* Subject treatment includes internal aortic cross-clamp or would have likely benefited from an internal aortic cross-clamp

Exclusion Criteria:

* Subject < 18 years of age
* Prisoner
* Evidence of cardiac, thoracic aortic, or great vessel injury identified in primary survey, FAST scan, and/or x-rays
* Any open/exsanguinating upper extremity wound

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: • All adult (age ≥ 18 years) trauma and acute care surgery patients treated with resuscitative AO (via open or endovascular means) in the acute phases after injury
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-29 (Actual); Primary Completion 2024-12-29 (Estimated); Study Completion 2024-12-29 (Estimated)

PRIMARY OUTCOMES:
Demographics | 01 July 2015 through 31st December 2024
  Age in years
Demographics- Gender | 01 July 2015 through 31st December 2024
  Male or Female
Demographics-Height | 01 July 2015 through 31st December 2024
  Height measured in Inches
Demographics- Weight | 01 July 2015 through 31st December 2024
  Weight measured in pounds
Injury Data | 01 July 2015 through 31st December 2024
  Mechanism classification - Penetrating, Blunt or Non-trauma Hemorrhage
Injury Mechanism Type | 01 July 2015 through 31st December 2024
  Gunshot wound, Motor vehicle accident, stab wound, fall
Body Region | 01 July 2015 through 31st December 2024
  Head/Neck, Chest, Abdomen, pelvis or Extremities

CONTACTS AND LOCATIONS:
Overall Officials: Conner McDaniel, M.D., Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No